CLINICAL TRIAL: NCT02550704
Title: Association Between High Faecal Calprotectin, Increased Intestinal Permeability and Visceral Hypersensitivity in Patients Suffering From Irritable Bowel Syndrome With Diarrhoea
Brief Title: Association Between High Faecal Calprotectin, Increased Intestinal Permeability and Visceral Hypersensitivity in IBS-D Patients
Acronym: SIIMPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Société Nationale Française de Gastroentérologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015/079/HP
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2021-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel syndrome; Intestinal permeability; Visceral hypersensitivity; Low grade inflammation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irritable Bowel Syndrome with diarrhea (Experimental): Colonoscopy with eleven biopsies in the left colon to assess intestinal permeability. Intestinal permeability is not routinely performed and is assessed in colonic biopsies (occludin, claudin and ZO-1 by western blot, qPCR and immunofluorescence)
  Interventions: Procedure: Colonoscopy with eleven biopsies in the left colon to assess intestinal permeability

INTERVENTIONS:
Procedure: Colonoscopy with eleven biopsies in the left colon to assess intestinal permeability — Eleven colonic biopsies are taken in the left colon during colonoscopy. Intestinal permeability is assessed by western blot, qPCR and immunofluorescence for claudin, occludin and ZO-1.

SUMMARY:
Visceral hypersensitivity, low grade inflammation and increased intestinal permeability are three main pathophysiological mechanisms involved in irritable bowel syndrome. The connexion between these abnormalities is not known. We hypothesis there is a link between them in IBS with diarrhoea.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional disorder which affect around 10% of the general population. Abdominal pain and discomfort are associated with transit disorders (diarrhea, constipation, alternating). IBS is defined by Rome III criteria.

For clinicians, IBS remains difficult to treat while its pathophysiology remains not completely understood. Visceral hypersensitivity, low grade inflammation and increased intestinal permeability are three abnormalities found in IBS patients. Visceral hypersensitivity is present in 60% of the patients, while intestinal permeability is increased in a subgroup of IBS with diarrhea. Low grade inflammation could be identify with faecal calprotectin dosage. The link between this three abnormalities is not clear.

The goal of our study is to describe the prevalence of these three abnormalities in IBS-Diarrhea population and to look for a correlation between low grade inflammation, visceral hypersensitivity, increased intestinal permeability and clinical phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* IBS-Diarrhoea according to Rome III criteria,
* Faecal calprotectin ≤200 µg/g in the last two months
* Effective contraception since 1 month for women in childbearing age

Exclusion Criteria:

* Patients with organic and/or inflammatory digestive disease
* IBS with constipation or alternating
* Treatment such as anti-inflammatory, probiotic in the last three months
* Patient with blood dyscrasia disorder known or identified , anticoagulant or antiplatelet treatments
* Small intestinal bacterial overgrowth (identified by a glucose breath test)
* Hypersensitivity to Normacol
* Severe renal failure
* Anal pathology (anal fissure, hemorrhoidal thrombosis)
* Pregnant or breastfeeding women
* Person with administrative or judicial decision or under legal protection measure
* Patient participating in another trial in the last two weeks
* Diet based in grapes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Occludin level expression in left colonic biopsies | day 1
  Occludin expression is measured using western blot (for proteins), Quantitative Real Time Polymerase Chain Reaction (q RT-PCR) (RNA) and IF (for localization)
Faecal calprotectin level | day 1
  Level is assessed on stool sample by ELISA kit in µg/g

SECONDARY OUTCOMES:
Claudin level expression in left colonic biopsies | day 1
  Claudin expression is measured using western blot (for proteins), q RT-PCR (for RNA) and IF (for localization)
Zonula Occludens (ZO)-1 level expression | day 1
  ZO-1 expression is measured using western blot (for proteins), q RT-PCR (for RNA) and IF (for localization)
Pression pain threshold by rectal barostat | day 1
  Pression pain threshold is measured in mmHg during rectal barostat.
Quality of life by GIQLI | day 1
  Evaluation of quality of life using the validated score : french version of the Gastrointestinal Quality of Life Index (GIQLI)
Abdominal symptoms | day 1
  Abdominal symptoms of IBS are assessed with IBS symptom severity scale.
Anxiety and depression level | day 1
  Anxiety and depression are assessed with the Hospital anxiety and depression scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Melchior, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France